CLINICAL TRIAL: NCT00353093
Title: Limited Versus Extended Ultrasonography for the Diagnosis of Clinically Symptomatic Deep Vein Thrombosis of the Lower Extremities. A Randomized Study
Brief Title: The ERASMUS Study: Limited vs Extended US for DVT Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 07/01
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 2005-07

CONDITIONS: Deep Vein Thrombosis of the Lower Extremities
Keywords: deep vein thrombosis,D-dimer,ultrasonography

INTERVENTIONS:
Procedure: Ultrasonography of the deep vein system of the legs

SUMMARY:
Currently, patients with suspected deep vein thrombosis (DVT) of the lower extremities receive the ultrasound investigation of their deep vein system, either by limited ultrasonography (ultrasonography confined to the proximal veins, repeating the test after one week in patients with positive D-dimer) or by extended ultrasonography (ultrasonography extented to the entire deep vein system of the legs). No study has directly compared the two strategies to assess their accuracy and safety. We plan to compare the accuracy and safety of the two strategies in a prospective randomized study addressing more than 2000 consecutive outpatients presenting with the clinical suspicion of DVT.

DETAILED DESCRIPTION:
All consecutive outpatients referred to the study center with clinically suspected deep vein thrombosis are potentially eligible for inclusion. Patients are excluded if they have a history of previous venous thromboembolism, have clinical suspicion of pulmonary embolism, have a life expectancy shorter than 3 months, have used therapeutic doses of unfractionated heparin, low molecular weight heparin or oral anticoagulants for more than 48 hours, have another indication for anticoagulant treatment, are pregnant, are aged less than 18 years, are inaccessible to follow-up, or refuse participation in the study.

Randomization Before randomization, patients are interviewed using a standardized questionnaire in order to collect information on risk factors for venous thrombosis, and the presence of several clinical signs and symptoms. Subsequently, they are randomized to the limited or the extended ultrasound strategy through computer generated lists, each of 100 patients arranged in balanced blocks of 10, specific for each center. The list is accessible only for a study nurse who informed the study physicians about group allocation once patients had provided informed consent.

Initial diagnostic workup Patients randomized to limited ultrasonography undergo compression ultrasonography, confining the investigation to the common femoral and the popliteal vein down to its trifurcation. In patients with normal findings D-dimer testing is performed, and they are subsequently managed according to its results: patients with normal D-dimer levels do not receive further investigation, while those with abnormal test are scheduled for repeat compression ultrasonography within one week.

Patients randomized to the extended ultrasonography receive first the evaluation of the proximal vein system, including the common femoral, the superficial femoral and the popliteal vein down its trifurcation. Then patients with compressible proximal veins undergo the extensive evaluation of the calf vein system, including the anterior tibial, posterior tibial and peroneal veins, and, if the deep veins were normal, also of the muscular (gastrocnemial and soleal) veins.

Limited ultrasonography and D-dimer The common femoral at the groin, and the popliteal vein down to its branching into the calf deep veins at the popliteal fossa, are examined in the transverse plane only, with a 7.5 MHz linear probe. The test results are categorized as normal (compressible veins) or abnormal (non compressible veins).

We use a rapid whole blood bedside D-dimer assay (SimpliRED® D-Dimer assay, AGEN Biomedical Ltd., Brisbane Australia). This assay is based on autologous red cell agglutination, using a chemical conjugate of a monoclonal antibody specific to human D-dimer (DD-3B6/22) linked to a monoclonal antibody which binds to the surface of human red blood cells (RAT-1C3/86) as active agent. The test can be performed either on capillary or on citrated venous blood. Agglutination occurs at D-dimer concentrations above 0.2 mg/L. The SimpliRED® results are categorized as normal, abnormal or non interpretable. The latter finding is categorized as abnormal.

Extended ultrasonography All veins are imaged along their length with a 7.5 MHz linear transducer. The proximal venous system is examined starting from the (common and superficial) femoral veins, which are scanned down to the distal part of the thigh, with the patient lying supine. Then, with the patient in the prone position the popliteal vein down to its trifurcation is evaluated. The calf veins are evaluated with the patient sitting with his/her legs hanging over the edge of the bed. Starting from the most proximal venous segments downwards, the anterior, posterior tibial and peroneal veins are visualized along their length, employing augmentation maneuvers (manual squeezing of the distal calf or of the foot) to enhance vessel visualization. The same approach is used to image the muscular veins. The only criterion to adjudicate a thrombosis involving the proximal system and the tibial and peroneal veins is the finding of a non compressible venous segment. As for the muscular veins, criteria for abnormal testing are incompressibility or the lack of spontaneous intraluminal color filling or reverse-flow color filling after augmentation maneuvers. All tests are performed by highly skilled physicians.

Follow-up All patients with an initial normal workup are discouraged from receiving antithrombotic drugs, and are scheduled for a clinical evaluation at three months. They are instructed to immediately contact the study centers should symptoms of venous thromboembolism become manifest in the meantime. In this case they undergo instrumental testing to confirm or refute the presence of the disease. Patients failing to attend the scheduled visit are contacted by telephone to assess their status, and invited to attend a clinical evaluation at the study centre.

Outcomes The primary outcomes of the study are: (1) the prevalence and location of venous thrombosis as shown by the initial diagnostic workup; (2) the rate of symptomatic venous thromboembolic events (including proximal vein thrombosis, isolated thrombosis of the tibial or peroneal veins in either leg, and pulmonary embolism) during three months of follow up in patients with an initially normal diagnostic workup. All suspected events are to be objectively evaluated as follows: ipsilateral or contralateral deep vein thrombosis is ruled in by abnormal compression ultrasonography or by the finding of an intraluminal filling defect on ascending venography, visible on two different projections; suspected pulmonary embolism is confirmed by an abnormal spiral computed tomography of the lung, by a high probability ventilation-perfusion lung scan, or by an abnormal pulmonary angiography. Fatal pulmonary embolism is adjudicated on the findings of autopsy, in case of sudden and otherwise inexplicable death, or on clinical grounds according to the opinion of an independent physician.

An independent and blind committee adjudicates all suspected thromboembolic events and all deaths occurring during the follow up based on all relevant documents and footage.

ELIGIBILITY:
Inclusion Criteria:

* outpatients with clinically suspected deep vein thrombosis of the lower extremities

Exclusion Criteria:

* history of previous venous thromboembolism
* clinical suspicion of pulmonary embolism
* life expectancy shorter than 3 months
* therapeutic doses of unfractionated heparin, low molecular weight heparin or oral anticoagulants for more than 48 hours
* another indication for anticoagulant treatment
* pregnancy
* age less than 18 years
* inaccessibility to follow-up
* refused participation in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2003-01; Study Completion 2005-07

PRIMARY OUTCOMES:
To assess(1) the prevalence and location of venous thrombosis
as shown by the initial diagnostic workup; (2) the rate of
symptomatic venous thromboembolic events (including proximal
vein thrombosis, isolated thrombosis of the tibial or peroneal
veins in either leg, and pulmonary embolism) during three months
of follow up in patients with an initially normal diagnostic workup.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Bernardi, MD, Principal Investigator — Department of Emergency and Accident Medicine, University Hospital of Padua

REFERENCES:
- [Derived] Bernardi E, Camporese G, Buller HR, Siragusa S, Imberti D, Berchio A, Ghirarduzzi A, Verlato F, Anastasio R, Prati C, Piccioli A, Pesavento R, Bova C, Maltempi P, Zanatta N, Cogo A, Cappelli R, Bucherini E, Cuppini S, Noventa F, Prandoni P; Erasmus Study Group. Serial 2-point ultrasonography plus D-dimer vs whole-leg color-coded Doppler ultrasonography for diagnosing suspected symptomatic deep vein thrombosis: a randomized controlled trial. JAMA. 2008 Oct 8;300(14):1653-9. doi: 10.1001/jama.300.14.1653. PMID 18840838